CLINICAL TRIAL: NCT03526744
Title: Dose Range Finding Study for Effects of Marine Protein Hydrolysate as Dietary Supplement in Elderly Active Subjects
Brief Title: Marine Protein Hydrolysate as Dietary Supplement in Elderly Part II
Acronym: MPH-DR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Møre og Romsdal HF (Other Government)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 2017/1795
Record Dates: First submitted 2018-04-26; First posted 2018-05-16 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Healthy Volunteers
Keywords: Dietary Supplements; Fish Proteins; Protein Hydrolysates; Aged

STUDY DESIGN:
Intervention Model Description: A simple open step-up design will be employed with no placebo control, but the sequence will be randomized. Both participant and investigator are blinded for the dose.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- marine protein hydrolysate 1234 (Experimental): Daily intake at breakfast of supplementary marine protein hydrolysate (MPH) equivalent to 10, 20, 30 or 40 mg per kg bodyweight during 1 week, followed by 3 similar cycles with other MPH dosages, with up to 7 days wash-out in between. Random sequence of arms.
  Interventions: Dietary Supplement: marine protein hydrolysate 1234
- marine protein hydrolysate 2134 (Experimental): Daily intake at breakfast of supplementary marine protein hydrolysate (MPH) equivalent to 10, 20, 30 or 40 mg per kg bodyweight during 1 week, followed by 3 similar cycles with other MPH dosages, with up to 7 days wash-out in between. Random sequence of arms.
  Interventions: Dietary Supplement: marine protein hydrolysate 2134
- marine protein hydrolysate 3124 (Experimental): Daily intake at breakfast of supplementary marine protein hydrolysate (MPH) equivalent to 10, 20, 30 or 40 mg per kg bodyweight during 1 week, followed by 3 similar cycles with other MPH dosages, with with up to 7 days-out in between. Random sequence of arms.
  Interventions: Dietary Supplement: marine protein hydrolysate 3124
- marine protein hydrolysate 4123 (Experimental): Daily intake at breakfast of supplementary marine protein hydrolysate (MPH) equivalent to 10, 20, 30 or 40 mg per kg bodyweight during 1 week, followed by 3 similar cycles with other MPH dosages, with up to 7 days wash-out in between. Random sequence of arms.
  Interventions: Dietary Supplement: marine protein hydrolysate 4123

INTERVENTIONS:
Dietary Supplement: marine protein hydrolysate 1234 — Dietary Supplement for e.g. in this order: MPH 1600 mg for 7 days, than 7 days wash-out. Dietary Supplement: MPH 800 mg for 7 days, than 7 days wash-out. Dietary Supplement: MPH 2400 mg for 7 days, than 7 days wash-out. Dietary Supplement: MPH 3200 mg for 7 days, than 7 days wash-out."
  Arms: marine protein hydrolysate 1234
Dietary Supplement: marine protein hydrolysate 2134 — Dietary Supplement for e.g. in this order: MPH 3200 mg for 7 days, than 7 days wash-out. Dietary Supplement: MPH 800 mg for 7 days, than 7 days wash-out. Dietary Supplement: MPH 2400 mg for 7 days, than 7 days wash-out. Dietary Supplement: MPH 1600 mg for 7 days, than 7 days wash-out."
  Arms: marine protein hydrolysate 2134
Dietary Supplement: marine protein hydrolysate 3124 — Dietary Supplement for e.g. in this order: MPH 2400 mg for 7 days, than 7 days wash-out. Dietary Supplement: MPH 3200 mg for 7 days, than 7 days wash-out. Dietary Supplement: MPH 1600 mg for 7 days, than 7 days wash-out. Dietary Supplement: MPH 800 mg for 7 days, than 7 days wash-out."
  Arms: marine protein hydrolysate 3124
Dietary Supplement: marine protein hydrolysate 4123 — Dietary Supplement for e.g. in this order: MPH 1600 mg for 7 days, than 7 days wash-out. Dietary Supplement: MPH 800 mg for 7 days, than 7 days wash-out. Dietary Supplement: MPH 3200 mg for 7 days, than 7 days wash-out. Dietary Supplement: MPH 2400 mg for 7 days, than 7 days wash-out."
  Arms: marine protein hydrolysate 4123

SUMMARY:
The aim of this study is to investigate the potential effect of different doses of MPH supplement on glucose metabolism, hunger and appetite hormones.

DETAILED DESCRIPTION:
The potential use of marine protein hydrolysates (MPH) as a supplement with similar or better health benefits than a regular white fish meal, can be regarded both cost-effective, environmental friendly and sustainable.

The aim of this study is to investigate the potential effect of increasing/different doses of MPH supplement on glucose metabolism, hunger and appetite hormones in healthy elderly, to provide a basis for the optimalization of the daily dose for further use of MPH in clinical study protocols in elderly patients with sarcopenia, other inflammatory conditions or abnormal glucose metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Body mass index (BMI) 20-30 kg/m2

Exclusion Criteria:

* Suspected allergies against fish or shellfish
* Low or unstable blood pressure
* Diabetes mellitus pharmacologically treated
* Chronic diseases or therapies that are likely to interfere with the evaluation of study results such as known inflammation or muscle loss
* Acute infections (may be reconsidered for inclusion at a later time)
* Substance misuse
* Inability or unwillingness to comply with the requirements of study procedures

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

PRIMARY OUTCOMES:
Glucose | A standardized meal, thereafter repeated measures every 20 minutes for 2 hours on day 7 in each intervention sequence
  Postprandial glucose (mmol/L) curve on day 7 in each sequence

SECONDARY OUTCOMES:
Insulin | After the standardized breakfast meal, repeated measure every 20 minutes for 2 hours, on day 7 in each intervention sequence
  Postprandial Insulin (mIE/L) - curve on day 7 in each sequence
Hormon 1 | At 6 different times point during a 2 hours period, on day 7 in each intervention sequence
  Glucagon like peptide 1 (GLP-1) pmol/l - curve, on day 7 in each sequence
Visual analogue scale (VAS) | Before breakfast on each study day (day 7 in each intervention sequence)
  Assessed by questionnaire VAS, scale from 0-10, where 0 is minimum score and 10 is the maximum score, reported e.g. as a total score of 7. The higher the reported value is the worse outcome.
KANE, symptom score | Two hours after breakfast on day 1 and 7 in each intervention sequence
  Assessed by questionaire KANE (Family name of an Author) , scale from 0-10, where 0 is minimum score and 10 is the maximum score, reported e.g. as a total score of 7. The higher the reported value is the worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dag Arne Lihaug Hoff, md phd, Study Director — Helse Møre & Romsdal HF, Ålesund Hospital
Locations (2):
- Norway (2):
  - Ålesund Hospital, Helse Møre og Romsdal HF, Ålesund
  - Haukeland University Hospital, Bergen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Jensen C, Dale HF, Hausken T, Lied E, Hatlebakk JG, Bronstad I, Lied GA, Hoff DAL. Supplementation with cod protein hydrolysate in older adults: a dose range cross-over study. J Nutr Sci. 2019 Dec 4;8:e40. doi: 10.1017/jns.2019.37. PMID 32042407
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC6984005/